CLINICAL TRIAL: NCT05947643
Title: Smell in COVID-19 and Efficacy of Nasal Theophylline 3
Brief Title: Smell in COVID-19 and Efficacy of Nasal Theophylline (SCENT 3)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 202209062
Record Dates: First submitted 2023-07-13; First posted 2023-07-17 (Actual); Results first posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: COVID-19
Keywords: Nasal Theophylline; Olfactory disfunction; Anosmia; Gustatory disorders; Dysgeusia
MeSH Terms: conditions — COVID-19; Anosmia; Dysgeusia | interventions — Theophylline

STUDY DESIGN:
Intervention Model Description: Single-site, double-blinded, placebo-controlled randomized clinical trial performed at a tertiary academic medical center.
Who Masked: Participant, Investigator
Masking Description: Double-blinded, meaning neither the subjects nor the investigators will be aware of the intervention received by any subject.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Theophylline (Experimental): Participants will dissolve the contents of the 400 mg theophylline capsules (experimental) into the sinus rinse bottle containing nasal saline.
  Interventions: Drug: theophylline
- Placebo (Placebo Comparator): Participant will dissolve the contents of the identical-appearing lactose capsules (control) into the sinus rinse bottle containing nasal saline.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: theophylline — capsules dissolved in intranasal irrigation
  Arms: Theophylline
Drug: Placebo — identical-appearing lactose capsules dissolved in intranasal irrigation
  Other Names: inactive medicine
  Arms: Placebo

SUMMARY:
The purpose of this Phase II trial is to test the effectiveness of intranasal theophylline irrigations for the treatment of COVID-19 related smell dysfunction. The investigators will compare the effect of theophylline nasal rinses versus placebo nasal rinses on smell symptoms. Participants will be asked to rinse their nose with a medication or placebo capsule dissolved in saltwater twice daily for 12 weeks and fill out surveys about smell before, during, and at the end of treatment.

This study will also be used to describe adverse effects related to intranasal theophylline irrigation.

DETAILED DESCRIPTION:
COVID-related olfactory dysfunction (OD) is a major symptom of infection with SARS-COV-2, affecting up to 80% of those with COVID-19. While research on the pathogenesis is ongoing, a significant subset is expected to suffer from long-term OD. The investigators seek to test intranasal theophylline nasal irrigation as a potential therapeutic option for treatment of COVID-related OD lasting over 3 months.

Theophylline has been shown to improve outcomes in post-viral OD in pilot studies, and initial data suggests therapeutic benefit in patients with post-COVID OD with minimal systemic absorption.

The primary hypothesis is that theophylline irrigation will be more effective than placebo saline irrigation for COVID-19 related OD symptoms. The use of intranasal theophylline will have minimal adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be recruited based on the following inclusion criteria:

  1. males and females ages 18 to 75 years
  2. located within or willing to travel to the state of Missouri or Illinois
  3. Olfactory dysfunction that has persisted for >3 months following suspected COVID-19 infection
  4. Baseline University of Pennsylvania Smell Identification Test (UPSIT) consistent with decreased olfactory function (<= 34 in women, <=33 in men). This test is a clinically validated 40-question forced-choice odor identification test where microencapsulated odorants on a strip are released by scratching.70 This will determine that patients have both subjectively and objectively diagnosed OD prior to undergoing treatment.
  5. Ability to read, write, and understand English and have access to email.

Exclusion Criteria:

* Individuals will not be allowed to participate in this study if they meet one or more of the following exclusion criteria:

  1. History of olfactory dysfunction prior to COVID-19 infection
  2. Any use of concomitant therapies specifically for the treatment of olfactory dysfunction
  3. Use of or participation in previous trials of intranasal theophylline.
  4. Known existence of nasal polyps, prior sinonasal, or anterior skull-based surgery
  5. Dependence on theophylline for comorbid conditions such as asthma and chronic obstructive pulmonary disease (COPD)
  6. History of an allergic reaction to theophylline or other methylxanthines
  7. History of neurodegenerative disease (ie. Alzheimer's dementia, Parkinson's disease, Lewy body dementia, frontotemporal dementia)
  8. Pregnant or breastfeeding mothers.
  9. Current use of medications with significant (≥40%) interactions with theophylline, which include cimetidine, ciprofloxacin, disulfiram, enoxacin, fluvoxamine, interferon- alpha, lithium, mexiletine, phenytoin, propafenone, propranolol, tacrine, thiabendazole, ticlopidine, and troleandomycin.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2022-11-22 (Actual); Primary Completion 2025-04-24 (Actual); Study Completion 2025-08-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jay F Piccirillo, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kaye R, Chang CWD, Kazahaya K, Brereton J, Denneny JC 3rd. COVID-19 Anosmia Reporting Tool: Initial Findings. Otolaryngol Head Neck Surg. 2020 Jul;163(1):132-134. doi: 10.1177/0194599820922992. Epub 2020 Apr 28. PMID 32340555
- [Background] Meng X, Deng Y, Dai Z, Meng Z. COVID-19 and anosmia: A review based on up-to-date knowledge. Am J Otolaryngol. 2020 Sep-Oct;41(5):102581. doi: 10.1016/j.amjoto.2020.102581. Epub 2020 Jun 2. PMID 32563019
- [Background] Whitcroft KL, Hummel T. Clinical Diagnosis and Current Management Strategies for Olfactory Dysfunction: A Review. JAMA Otolaryngol Head Neck Surg. 2019 Sep 1;145(9):846-853. doi: 10.1001/jamaoto.2019.1728. PMID 31318413
- [Background] Dong E, Ratcliff J, Goyea TD, Katz A, Lau R, Ng TK, Garcia B, Bolt E, Prata S, Zhang D, Murray RC, Blake MR, Du H, Ganjkhanloo F, Ahmadi F, Williams J, Choudhury S, Gardner LM. The Johns Hopkins University Center for Systems Science and Engineering COVID-19 Dashboard: data collection process, challenges faced, and lessons learned. Lancet Infect Dis. 2022 Dec;22(12):e370-e376. doi: 10.1016/S1473-3099(22)00434-0. Epub 2022 Aug 31. PMID 36057267
- [Background] Menni C, Valdes AM, Polidori L, Antonelli M, Penamakuri S, Nogal A, Louca P, May A, Figueiredo JC, Hu C, Molteni E, Canas L, Osterdahl MF, Modat M, Sudre CH, Fox B, Hammers A, Wolf J, Capdevila J, Chan AT, David SP, Steves CJ, Ourselin S, Spector TD. Symptom prevalence, duration, and risk of hospital admission in individuals infected with SARS-CoV-2 during periods of omicron and delta variant dominance: a prospective observational study from the ZOE COVID Study. Lancet. 2022 Apr 23;399(10335):1618-1624. doi: 10.1016/S0140-6736(22)00327-0. Epub 2022 Apr 7. PMID 35397851
- [Background] Chen M, Pekosz A, Villano JS, Shen W, Zhou R, Kulaga H, Li Z, Smith A, Gurung A, Beck SE, Witwer KW, Mankowski JL, Ramanathan M Jr, Rowan NR, Lane AP. Evolution of nasal and olfactory infection characteristics of SARS-CoV-2 variants. J Clin Invest. 2024 Mar 14;134(8):e174439. doi: 10.1172/JCI174439. PMID 38483537
- [Background] Sedaghat AR, Gengler I, Speth MM. Olfactory Dysfunction: A Highly Prevalent Symptom of COVID-19 With Public Health Significance. Otolaryngol Head Neck Surg. 2020 Jul;163(1):12-15. doi: 10.1177/0194599820926464. Epub 2020 May 5. PMID 32366160
- [Background] Moein ST, Hashemian SM, Mansourafshar B, Khorram-Tousi A, Tabarsi P, Doty RL. Smell dysfunction: a biomarker for COVID-19. Int Forum Allergy Rhinol. 2020 Aug;10(8):944-950. doi: 10.1002/alr.22587. Epub 2020 Jun 18. PMID 32301284
- [Background] Menni C, Sudre CH, Steves CJ, Ourselin S, Spector TD. Quantifying additional COVID-19 symptoms will save lives. Lancet. 2020 Jun 20;395(10241):e107-e108. doi: 10.1016/S0140-6736(20)31281-2. Epub 2020 Jun 4. No abstract available. PMID 32505221
- [Background] Carfi A, Bernabei R, Landi F; Gemelli Against COVID-19 Post-Acute Care Study Group. Persistent Symptoms in Patients After Acute COVID-19. JAMA. 2020 Aug 11;324(6):603-605. doi: 10.1001/jama.2020.12603. PMID 32644129
- [Background] Tan BKJ, Han R, Zhao JJ, Tan NKW, Quah ESH, Tan CJ, Chan YH, Teo NWY, Charn TC, See A, Xu S, Chapurin N, Chandra RK, Chowdhury N, Butowt R, von Bartheld CS, Kumar BN, Hopkins C, Toh ST. Prognosis and persistence of smell and taste dysfunction in patients with covid-19: meta-analysis with parametric cure modelling of recovery curves. BMJ. 2022 Jul 27;378:e069503. doi: 10.1136/bmj-2021-069503. PMID 35896188
- [Background] Whitcroft KL, Hummel T. Olfactory Dysfunction in COVID-19: Diagnosis and Management. JAMA. 2020 Jun 23;323(24):2512-2514. doi: 10.1001/jama.2020.8391. No abstract available. PMID 32432682
- [Background] Catton G, Gardner A. COVID-19 Induced Taste Dysfunction and Recovery: Association with Smell Dysfunction and Oral Health Behaviour. Medicina (Kaunas). 2022 May 26;58(6):715. doi: 10.3390/medicina58060715. PMID 35743978
- [Background] Sungnak W, Huang N, Becavin C, Berg M, Queen R, Litvinukova M, Talavera-Lopez C, Maatz H, Reichart D, Sampaziotis F, Worlock KB, Yoshida M, Barnes JL; HCA Lung Biological Network. SARS-CoV-2 entry factors are highly expressed in nasal epithelial cells together with innate immune genes. Nat Med. 2020 May;26(5):681-687. doi: 10.1038/s41591-020-0868-6. Epub 2020 Apr 23. PMID 32327758
- [Background] Rockx B, Kuiken T, Herfst S, Bestebroer T, Lamers MM, Oude Munnink BB, de Meulder D, van Amerongen G, van den Brand J, Okba NMA, Schipper D, van Run P, Leijten L, Sikkema R, Verschoor E, Verstrepen B, Bogers W, Langermans J, Drosten C, Fentener van Vlissingen M, Fouchier R, de Swart R, Koopmans M, Haagmans BL. Comparative pathogenesis of COVID-19, MERS, and SARS in a nonhuman primate model. Science. 2020 May 29;368(6494):1012-1015. doi: 10.1126/science.abb7314. Epub 2020 Apr 17. PMID 32303590
- [Background] Zou L, Ruan F, Huang M, Liang L, Huang H, Hong Z, Yu J, Kang M, Song Y, Xia J, Guo Q, Song T, He J, Yen HL, Peiris M, Wu J. SARS-CoV-2 Viral Load in Upper Respiratory Specimens of Infected Patients. N Engl J Med. 2020 Mar 19;382(12):1177-1179. doi: 10.1056/NEJMc2001737. Epub 2020 Feb 19. No abstract available. PMID 32074444
- [Background] Baig AM, Khaleeq A, Ali U, Syeda H. Evidence of the COVID-19 Virus Targeting the CNS: Tissue Distribution, Host-Virus Interaction, and Proposed Neurotropic Mechanisms. ACS Chem Neurosci. 2020 Apr 1;11(7):995-998. doi: 10.1021/acschemneuro.0c00122. Epub 2020 Mar 13. PMID 32167747
- [Background] Brann DH, Tsukahara T, Weinreb C, Lipovsek M, Van den Berge K, Gong B, Chance R, Macaulay IC, Chou HJ, Fletcher RB, Das D, Street K, de Bezieux HR, Choi YG, Risso D, Dudoit S, Purdom E, Mill J, Hachem RA, Matsunami H, Logan DW, Goldstein BJ, Grubb MS, Ngai J, Datta SR. Non-neuronal expression of SARS-CoV-2 entry genes in the olfactory system suggests mechanisms underlying COVID-19-associated anosmia. Sci Adv. 2020 Jul 31;6(31):eabc5801. doi: 10.1126/sciadv.abc5801. Epub 2020 Jul 24. PMID 32937591
- [Background] Morbini P, Benazzo M, Verga L, Pagella FG, Mojoli F, Bruno R, Marena C. Ultrastructural Evidence of Direct Viral Damage to the Olfactory Complex in Patients Testing Positive for SARS-CoV-2. JAMA Otolaryngol Head Neck Surg. 2020 Oct 1;146(10):972-973. doi: 10.1001/jamaoto.2020.2366. No abstract available. PMID 32790835
- [Background] Politi LS, Salsano E, Grimaldi M. Magnetic Resonance Imaging Alteration of the Brain in a Patient With Coronavirus Disease 2019 (COVID-19) and Anosmia. JAMA Neurol. 2020 Aug 1;77(8):1028-1029. doi: 10.1001/jamaneurol.2020.2125. No abstract available. PMID 32469400
- [Background] Pekala K, Chandra RK, Turner JH. Efficacy of olfactory training in patients with olfactory loss: a systematic review and meta-analysis. Int Forum Allergy Rhinol. 2016 Mar;6(3):299-307. doi: 10.1002/alr.21669. Epub 2015 Dec 1. PMID 26624966
- [Background] Wilson DA, Best AR, Sullivan RM. Plasticity in the olfactory system: lessons for the neurobiology of memory. Neuroscientist. 2004 Dec;10(6):513-24. doi: 10.1177/1073858404267048. PMID 15534037
- [Background] Kollndorfer K, Kowalczyk K, Hoche E, Mueller CA, Pollak M, Trattnig S, Schopf V. Recovery of olfactory function induces neuroplasticity effects in patients with smell loss. Neural Plast. 2014;2014:140419. doi: 10.1155/2014/140419. Epub 2014 Dec 3. PMID 25544900
- [Background] Hoffman HJ, Rawal S, Li CM, Duffy VB. New chemosensory component in the U.S. National Health and Nutrition Examination Survey (NHANES): first-year results for measured olfactory dysfunction. Rev Endocr Metab Disord. 2016 Jun;17(2):221-40. doi: 10.1007/s11154-016-9364-1. PMID 27287364
- [Background] Liu B, Luo Z, Pinto JM, Shiroma EJ, Tranah GJ, Wirdefeldt K, Fang F, Harris TB, Chen H. Relationship Between Poor Olfaction and Mortality Among Community-Dwelling Older Adults: A Cohort Study. Ann Intern Med. 2019 May 21;170(10):673-681. doi: 10.7326/M18-0775. Epub 2019 Apr 30. PMID 31035288
- [Background] Pinto JM, Wroblewski KE, Kern DW, Schumm LP, McClintock MK. Olfactory dysfunction predicts 5-year mortality in older adults. PLoS One. 2014 Oct 1;9(10):e107541. doi: 10.1371/journal.pone.0107541. eCollection 2014. PMID 25271633
- [Background] Van Regemorter V, Hummel T, Rosenzweig F, Mouraux A, Rombaux P, Huart C. Mechanisms Linking Olfactory Impairment and Risk of Mortality. Front Neurosci. 2020 Feb 21;14:140. doi: 10.3389/fnins.2020.00140. eCollection 2020. PMID 32153360
- [Background] Soler ZM, Patel ZM, Turner JH, Holbrook EH. A primer on viral-associated olfactory loss in the era of COVID-19. Int Forum Allergy Rhinol. 2020 Jul;10(7):814-820. doi: 10.1002/alr.22578. Epub 2020 Jun 1. PMID 32271490
- [Background] Bitter T, Gudziol H, Burmeister HP, Mentzel HJ, Guntinas-Lichius O, Gaser C. Anosmia leads to a loss of gray matter in cortical brain areas. Chem Senses. 2010 Jun;35(5):407-15. doi: 10.1093/chemse/bjq028. Epub 2010 Mar 15. PMID 20231262
- [Background] Murphy C, Schubert CR, Cruickshanks KJ, Klein BE, Klein R, Nondahl DM. Prevalence of olfactory impairment in older adults. JAMA. 2002 Nov 13;288(18):2307-12. doi: 10.1001/jama.288.18.2307. PMID 12425708
- [Background] Cho SH. Clinical Diagnosis and Treatment of Olfactory Dysfunction. Hanyang Med Rev. 2014;34(3):107-115.
- [Background] Schiffman SS, Warwick ZS. Flavor enhancement of foods for the elderly can reverse anorexia. Neurobiol Aging. 1988 Jan-Feb;9(1):24-6. doi: 10.1016/s0197-4580(88)80009-5. PMID 3164095
- [Background] Hendriks AP. Olfactory dysfunction. Rhinology. 1988 Dec;26(4):229-51. PMID 3070710
- [Background] Reden J, Mueller A, Mueller C, Konstantinidis I, Frasnelli J, Landis BN, Hummel T. Recovery of olfactory function following closed head injury or infections of the upper respiratory tract. Arch Otolaryngol Head Neck Surg. 2006 Mar;132(3):265-9. doi: 10.1001/archotol.132.3.265. PMID 16549746
- [Background] RECOVERY Collaborative Group; Horby P, Lim WS, Emberson JR, Mafham M, Bell JL, Linsell L, Staplin N, Brightling C, Ustianowski A, Elmahi E, Prudon B, Green C, Felton T, Chadwick D, Rege K, Fegan C, Chappell LC, Faust SN, Jaki T, Jeffery K, Montgomery A, Rowan K, Juszczak E, Baillie JK, Haynes R, Landray MJ. Dexamethasone in Hospitalized Patients with Covid-19. N Engl J Med. 2021 Feb 25;384(8):693-704. doi: 10.1056/NEJMoa2021436. Epub 2020 Jul 17. PMID 32678530
- [Background] Sorokowska A, Drechsler E, Karwowski M, Hummel T. Effects of olfactory training: a meta-analysis. Rhinology. 2017 Mar 1;55(1):17-26. doi: 10.4193/Rhino16.195. PMID 28040824
- [Background] Konstantinidis I, Tsakiropoulou E, Bekiaridou P, Kazantzidou C, Constantinidis J. Use of olfactory training in post-traumatic and postinfectious olfactory dysfunction. Laryngoscope. 2013 Dec;123(12):E85-90. doi: 10.1002/lary.24390. Epub 2013 Oct 4. PMID 24114690
- [Background] Konstantinidis I, Tsakiropoulou E, Constantinidis J. Long term effects of olfactory training in patients with post-infectious olfactory loss. Rhinology. 2016 Jun;54(2):170-5. doi: 10.4193/Rhino15.264. PMID 27017331
- [Background] Hura N, Xie DX, Choby GW, Schlosser RJ, Orlov CP, Seal SM, Rowan NR. Treatment of post-viral olfactory dysfunction: an evidence-based review with recommendations. Int Forum Allergy Rhinol. 2020 Sep;10(9):1065-1086. doi: 10.1002/alr.22624. Epub 2020 Jun 25. PMID 32567798
- [Background] Cerebrolycin for Treatment of Covid-related Anosmia and Ageusia.
- [Background] Moon C, Simpson PJ, Tu Y, Cho H, Ronnett GV. Regulation of intracellular cyclic GMP levels in olfactory sensory neurons. J Neurochem. 2005 Oct;95(1):200-9. doi: 10.1111/j.1471-4159.2005.03356.x. PMID 16181424
- [Background] Pace U, Hanski E, Salomon Y, Lancet D. Odorant-sensitive adenylate cyclase may mediate olfactory reception. Nature. 1985 Jul 18-24;316(6025):255-8. doi: 10.1038/316255a0. PMID 3927168
- [Background] Barnes PJ. Theophylline. Pharmaceuticals (Basel). 2010 Mar 18;3(3):725-747. doi: 10.3390/ph3030725. PMID 27713276
- [Background] Ronnett GV, Parfitt DJ, Hester LD, Snyder SH. Odorant-sensitive adenylate cyclase: rapid, potent activation and desensitization in primary olfactory neuronal cultures. Proc Natl Acad Sci U S A. 1991 Mar 15;88(6):2366-9. doi: 10.1073/pnas.88.6.2366. PMID 2006174
- [Background] Anholt RR. Molecular neurobiology of olfaction. Crit Rev Neurobiol. 1993;7(1):1-22. PMID 8467526
- [Background] Neumann S, Bradke F, Tessier-Lavigne M, Basbaum AI. Regeneration of sensory axons within the injured spinal cord induced by intraganglionic cAMP elevation. Neuron. 2002 Jun 13;34(6):885-93. doi: 10.1016/s0896-6273(02)00702-x. PMID 12086637
- [Background] Henkin RI, Velicu I. cAMP and cGMP in nasal mucus: relationships to taste and smell dysfunction, gender and age. Clin Invest Med. 2008;31(2):E71-7. doi: 10.25011/cim.v31i2.3366. PMID 18377763
- [Background] Henkin RI, Velicu I. cAMP and cGMP in nasal mucus related to severity of smell loss in patients with smell dysfunction. Clin Invest Med. 2008;31(2):E78-84. doi: 10.25011/cim.v31i2.3367. PMID 18377764
- [Background] Henkin RI, Velicu I, Schmidt L. An open-label controlled trial of theophylline for treatment of patients with hyposmia. Am J Med Sci. 2009 Jun;337(6):396-406. doi: 10.1097/MAJ.0b013e3181914a97. PMID 19359985
- [Background] Levy LM, Henkin RI, Lin CS, Hutter A, Schellinger D. Increased brain activation in response to odors in patients with hyposmia after theophylline treatment demonstrated by fMRI. J Comput Assist Tomogr. 1998 Sep-Oct;22(5):760-70. doi: 10.1097/00004728-199809000-00019. PMID 9754114
- [Background] AlAjmi MF, Azhar A, Owais M, Rashid S, Hasan S, Hussain A, Rehman MT. Antiviral potential of some novel structural analogs of standard drugs repurposed for the treatment of COVID-19. J Biomol Struct Dyn. 2021 Oct;39(17):6676-6688. doi: 10.1080/07391102.2020.1799865. Epub 2020 Jul 30. PMID 32729392
- [Background] Elzupir AO. Caffeine and caffeine-containing pharmaceuticals as promising inhibitors for 3-chymotrypsin-like protease of SARS-CoV-2. J Biomol Struct Dyn. 2022 Mar;40(5):2113-2120. doi: 10.1080/07391102.2020.1835732. Epub 2020 Oct 23. PMID 33094705
- [Background] Tomita K, Chikumi H, Tokuyasu H, Yajima H, Hitsuda Y, Matsumoto Y, Sasaki T. Functional assay of NF-kappaB translocation into nuclei by laser scanning cytometry: inhibitory effect by dexamethasone or theophylline. Naunyn Schmiedebergs Arch Pharmacol. 1999 Apr;359(4):249-55. doi: 10.1007/pl00005349. PMID 10344522
- [Background] Henkin RI, Schultz M, Minnick-Poppe L. Intranasal theophylline treatment of hyposmia and hypogeusia: a pilot study. Arch Otolaryngol Head Neck Surg. 2012 Nov;138(11):1064-70. doi: 10.1001/2013.jamaoto.342. PMID 23165381
- [Background] Goldstein MF, Hilditch GJ, Frankel I, Chambers L, Dvorin DJ, Belecanech G. Intra-Nasal Theophylline for the Treatment of Chronic Anosmia and Hyposmia. Journal of Allergy and Clinical Immunology. 2017;139(2):AB252.
- [Background] Gupta S, Lee JJ, Perrin A, Khan A, Smith HJ, Farrell N, Kallogjeri D, Piccirillo JF. Efficacy and Safety of Saline Nasal Irrigation Plus Theophylline for Treatment of COVID-19-Related Olfactory Dysfunction: The SCENT2 Phase 2 Randomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2022 Sep 1;148(9):830-837. doi: 10.1001/jamaoto.2022.1573. PMID 35797024
- [Background] Dunlop BW, Gray J, Rapaport MH. Transdiagnostic Clinical Global Impression Scoring for Routine Clinical Settings. Behav Sci (Basel). 2017 Jun 27;7(3):40. doi: 10.3390/bs7030040. PMID 28653978
- [Background] Barnes PJ. Theophylline in chronic obstructive pulmonary disease: new horizons. Proc Am Thorac Soc. 2005;2(4):334-9; discussion 340-1. doi: 10.1513/pats.200504-024SR. PMID 16267358
- [Background] Tzelepis GE, Bascom AT, Safwan Badr M, Goshgarian HG. Effects of theophylline on pulmonary function in patients with traumatic tetraplegia. J Spinal Cord Med. 2006;29(3):227-33. doi: 10.1080/10790268.2006.11753878. PMID 16859226
- [Background] Yu TJ, Liu YC, Chu CM, Hu HC, Kao KC. Effects of theophylline therapy on respiratory muscle strength in patients with prolonged mechanical ventilation: A retrospective cohort study. Medicine (Baltimore). 2019 Jan;98(2):e13982. doi: 10.1097/MD.0000000000013982. PMID 30633180
- [Background] McKay SE, Howie CA, Thomson AH, Whiting B, Addis GJ. Value of theophylline treatment in patients handicapped by chronic obstructive lung disease. Thorax. 1993 Mar;48(3):227-32. doi: 10.1136/thx.48.3.227. PMID 8497820
- [Background] Hosein W, Henkin RI. Therapeutic diminution of Interleukin-10 with intranasal theophylline administration in hyposmic patients. Am J Otolaryngol. 2022 Mar-Apr;43(2):103375. doi: 10.1016/j.amjoto.2022.103375. Epub 2022 Jan 28. PMID 35124402
- [Background] Lee JJ, Peterson AM, Kallogjeri D, Jiramongkolchai P, Kukuljan S, Schneider JS, Klatt-Cromwell CN, Drescher AJ, Brunworth JD, Piccirillo JF. Smell Changes and Efficacy of Nasal Theophylline (SCENT) irrigation: A randomized controlled trial for treatment of post-viral olfactory dysfunction. Am J Otolaryngol. 2022 Mar-Apr;43(2):103299. doi: 10.1016/j.amjoto.2021.103299. Epub 2021 Dec 3. PMID 34894449
- [Background] Lee JJ, Gupta S, Kallogjeri D, Piccirillo JF. Safety of High-Dose Nasal Theophylline Irrigation in the Treatment of Postviral Olfactory Dysfunction: A Dose-Escalation Study. JAMA Otolaryngol Head Neck Surg. 2022 Sep 1;148(9):885-886. doi: 10.1001/jamaoto.2022.1574. PMID 35797023
- [Background] Doty RL, Shaman P, Dann M. Development of the University of Pennsylvania Smell Identification Test: a standardized microencapsulated test of olfactory function. Physiol Behav. 1984 Mar;32(3):489-502. doi: 10.1016/0031-9384(84)90269-5. PMID 6463130
- [Background] Theophylline in Dextrose [package insert]. Lake Forest, IL: Hospira, INC;2008
- See also: Anosmia Rehabilitation in Patients Post Coronavirus Disease (COVID 19). — https://ClinicalTrials.gov/show/NCT04374474.
- See also: COVID-19 Anosmia Study. — https://ClinicalTrials.gov/show/NCT04495816.
- See also: Corticosteroid Nasal Spray in COVID-19 Anosmia. — https://ClinicalTrials.gov/show/NCT04484493.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Per protocol the study plans to enroll 240 patients to account for a 20% dropout rate, aiming to have 200 evaluable participants for the trial.
  Reported are 77 randomized patients.
Period: Overall Study
Arm/Group | Theophylline | Placebo
Started | 39 | 38
Completed | 21 | 27
Not Completed | 18 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Theophylline | Placebo | Total
Number analyzed (Participants) | 39 | 38 | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (14) | 49 (13) | 48 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 26 | 56
  Male | 9 | 12 | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaskan Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  Hispanic or Latino | 1 | 0 | 1
  Native Hawaiian or pacific Islander | 0 | 0 | 0
  White | 18 | 25 | 43
  Asian and White | 0 | 1 | 1
Parosmia [Count of Participants; unit: Participants]
  Yes | 28 | 29 | 57
  No | 11 | 9 | 20
Phantosmia [Count of Participants; unit: Participants]
  Yes | 17 | 17 | 34
  No | 22 | 21 | 43
The University of Pennsylvania Smell Identification Test [Median (Full Range); unit: score on a scale (0-40)] — The University of Pennsylvania Smell Identification Test (UPSIT) is a clinically validated, 40-question forced-choice odor identification test used to objectively assess olfactory function. UPSIT scores help determine the presence and severity of olfactory dysfunction, with specific cutoff values indicating decreased olfactory function (≤34 for women, ≤33 for men).
  Higher scores indicate better olfactory function, and lower scores reflect greater olfactory dysfunction.
  score on a scale (0-40) | 25 [5 to 34] | 28 [7 to 34] | 25 [5 to 34]
The Olfactory Dysfunction Outcomes Rating [Median (Full Range); unit: score on a scale 0-112] — The The Olfactory Dysfunction Outcomes Rating (ODOR) scale consists of 28 questions, each addressing a specific aspect of how olfactory dysfunction impacts a person's life.
  Each question is typically answered on a Likert scale, ranging from 0 (no difficulty or very rarely bothered) to 4 (complete difficulty or very frequently bothered).
  The scores for all 28 items are summed to obtain a total score, which can range from 0 to 112 points.
  score on a scale 0-112 | 52 [0 to 105] | 47 [14 to 89] | 49 [0 to 105]
Clinical Global Impression of Severity of Smell Loss [Count of Participants; unit: Participants]
  Absent | 7 | 6 | 13
  Poor | 25 | 21 | 46
  Fair | 5 | 9 | 14
  Good | 0 | 1 | 1
  Very Good | 0 | 1 | 1
  Excellent | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Clinical Global Impression - Improvement Scale
Description: The Clinical Global Impression-Improvement scale (CGI-I) is a subjective rating scale used to measure changes in a patient's condition over time. It ranges from 1 to 7, where 1 means "Very Much Improved," 2 means "Much Improved," 3 means "Minimally Improved," 4 means "No Change," 5 means "Minimally Worse," 6 means "Much Worse," and 7 means "Very Much Worsened." In this study, participants reporting scores of 1, 2, or 3 on the CGI-I are considered responders to treatment. The primary analysis will compare the proportion of responders between the theophylline and placebo groups assessing both within-subject changes over time and between-group differences.
  We will measure the response rate defined as the number of participants self-reporting minimal change or larger in the Clinical Global Impression Scale (CGI) scale, divided by the number of participants in each group.The main comparison will be focused on changes at 12-weeks
Time Frame: week 12
Measure: Count of Participants; unit: Participants
Arm/Group | Theophylline | Placebo
Number analyzed (Participants) | 21 | 27
Participants | 9 | 9

2. Secondary Outcome: Olfactory Dysfunction Outcomes Rating
Description: Olfactory Dysfunction Outcomes Rating (ODOR) is a disease-specific questionnaire that assesses for physical, functional, and emotional limitations in participants with olfactory dysfunction of any etiology. The instrument contains 28 total items with each scored on a 5-point Likert scale from 0 to 4.
  Total score ranges from 0 to 112. Higher scores indicate higher degree of dysfunction and limitation.
Time Frame: 6 weeks and 12 week
Measure: Mean (95% Confidence Interval); unit: score on a scale (0-112)
Arm/Group | Theophylline | Placebo
Number analyzed (Participants) | 21 | 27
score on a scale (0-112)
  6 weeks | 43.38 [34.35 to 52.41] | 45.96 [38.21 to 53.72]
  12 weeks | 43.94 [35.08 to 52.80] | 45.26 [37.33 to 53.18]

3. Secondary Outcome: Assessment of Adherence
Description: Participants will be contacted to report the number of irrigations completed over the prior 7 days out of a possible 14.
  Participants report their compliance with the twice-daily nasal irrigations through self-reported measures in REDCap surveys, including how many rinses they have completed.
  The measure count represents the self-reported compliance with twice daily irrigations.
Time Frame: 12 weeks
Measure: Number; unit: participants
Arm/Group | Theophylline | Placebo
Number analyzed (Participants) | 29 | 32
participants
  6 days | 1 | 1
  8 days | 1 | 0
  10 days | 1 | 1
  11 days | 1 | 0
  12 days | 5 | 1
  13 days | 2 | 4
  14 days | 18 | 25

4. Secondary Outcome: Assessment of Blind
Description: The assessment of the blind in this study involves contacting participants within the first 3 weeks after starting nasal irrigations and asking them which treatment arm they believe they were assigned to-either "theophylline and nasal saline irrigation" or "nasal saline irrigation alone."
  The numbers reported represent how many participants correctly guessed an arm in which they were assigned to.
Time Frame: within first 3 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Theophylline | Placebo
Number analyzed (Participants) | 39 | 38
Participants | 20 | 26

5. Secondary Outcome: Adverse Effects
Description: Patients will be asked to report any adverse effects they experience at any time during the 12-week study period.
  An adverse event in this study refers to any undesirable or unintended medical occurrence experienced by a participant during the trial, which may or may not be related to the use of intranasal theophylline.
Time Frame: up to 12 weeks
Measure: Number; unit: participants
Arm/Group | Theophylline | Placebo
Number analyzed (Participants) | 39 | 38
participants
  Mild nose bleed | 1 | 0
  Dry nose noted and blood-tinged nasal discharge | 1 | 0
  Small amount of epistaxis and cold during the first week. | 1 | 0
  Upper respiratory infection and sleep disturbing cough | 1 | 0
  Little hard red bumps inside and outside of nose. | 0 | 1
  Migraine | 0 | 1
  Participant developed a sinus infection | 0 | 3
  Patient developed nausea, vomiting, and diarrhea | 0 | 1
  Nasal soreness | 0 | 1
  Urine in blood | 0 | 1

ADVERSE EVENTS:
Time Frame: Adverse event data will be collected throughout the entire 12-week study period. Specifically, participants will be asked about adverse events during phone check-ins at weeks 3, 6, 9, and 12. Additionally, participants can report adverse events at any time by contacting the study team via phone or pager, who are available 24/7 during the trial.
Description: Common systemic adverse effects of theophylline include headache, nausea, vomiting, tremors, insomnia, lightheadedness, and restlessness, while serious effects can include tachyarrhythmias, atrial fibrillation, Stevens-Johnson syndrome, intracranial hemorrhage, and seizure. However, intranasal theophylline has shown minimal adverse effects and negligible systemic absorption in prior studies.
Arm/Group | Theophylline | Placebo
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/38
Other Adverse Events (participants affected / at risk) | 4/39 | 8/38
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Theophylline (N=39) | Placebo (N=38)
mid nose bleed (General disorders) | 1 (1) | 0 (0)
Dry nose noted and blood tingled nasal discharge (General disorders) | 1 (1) | 0 (0)
Small amount of epistaxis and cold during the first week (General disorders) | 1 (1) | 0 (0)
Upper respiratory of infection and sleep disturbing cough (General disorders) | 1 (1) | 0 (0)
Little hard red bumps inside and outside of nose (General disorders) | 0 (0) | 1 (1)
Migraine (General disorders) | 0 (0) | 1 (1)
Participants developed a sinus infection (General disorders) | 0 (0) | 3 (3)
Patient developed nausea, vomiting and diarrhea (General disorders) | 0 (0) | 1 (1)
Nasal soreness (General disorders) | 0 (0) | 1 (1)
Urine in blood (General disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The exact pathogenesis of COVID-related anosmia remains unclear, complicating targeted treatment development. Prior treatments like corticosteroids and olfactory training have shown limited or variable efficacy, and no gold standard exists.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-06): https://cdn.clinicaltrials.gov/large-docs/43/NCT05947643/Prot_SAP_000.pdf